CLINICAL TRIAL: NCT05017038
Title: The Role of Social and Territorial Inequalities in the Management and Prognosis of Multiple Sclerosis - Longitudinal Observational Study - INESEP
Brief Title: The Role of Social and Territorial Inequalities in the Management and Prognosis of Multiple Sclerosis
Acronym: INESEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02739-48
Record Dates: First submitted 2021-08-19; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis; Social and Territorial Inequalities
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although the majority of the French population is covered by social security, the effects of social inequalities on health are still very visible and are even increasing in France and in Europe. Thus, according to INSEE, excess mortality is observed among the most disadvantaged populations. Similarly, the prevalence of certain chronic diseases in France and Europe, particularly cardiovascular diseases, is linked to social inequalities and excess morbidity can be observed in the most disadvantaged populations.

In addition to social inequalities, which refer to disparities in health levels according to social category, there are the effects of territorial inequalities. In France, there are geographical areas of excess mortality, which essentially correspond to areas far from urban centers. Similarly, there are major geographical differences in terms of medical supply and equipment, and the distance between patients and health centers is a direct obstacle to the use of the health care network.

The underlying explanations for social inequalities in health are multiple. While it is likely that difficulties in accessing and using care play a role, it is also possible that they are due to differences in exposure to certain environmental (e.g. pollution) or individual (e.g. smoking) risk factors. But it is also possible that the causal relationship is the opposite and that diseases create or reveal social inequalities.

For multiple sclerosis (MS) the impact of social and territorial inequalities is more debated. Indeed, with regard to the relationship between disease prevalence and social inequalities, a recent literature review found 21 separate studies on the subject, of which 13 failed to show a link between socioeconomic status and MS risk, 5 concluded that there was an increased risk of MS in advantaged populations and 3 concluded that there was an increased risk of MS in disadvantaged populations. There are plausible pathophysiological explanations for either direction of the relationship, but the question remains open.

To our knowledge, the link between MS prognosis and social inequalities has been little studied, as disadvantaged populations are more often exposed to the poor prognostic factor of smoking [6-8], the hypothesis of a negative prognostic role of social inequalities remains plausible. Similarly, the current consensus is that the diagnosis and treatment of MS should be as early as possible [9,10] in order to preserve brain capital. Easy access to a neurologist and MRI are therefore potentially prognostic factors for MS in relation to territorial inequalities. It should be noted that the link between social and geographical inequalities and a potential delay in treatment has not been demonstrated in France in the case of cancer, but it is possible that the importance of the means implemented in the fight against cancer erases these effects. In MS, a study showed a link between delay in starting a second disease-modifying therapy and socio-economic status.

While the causal link between MS and socio-professional status has not yet been demonstrated, the socio-economic impact of MS has been measured. In particular, it has been shown that having MS is associated with an increased risk of unemployment and/or early retirement.

The primary objective of our study is to determine whether delay in treatment, as a marker of difficulties in access to care in MS, is associated with social and territorial inequalities in MS. Secondary objectives will be to explore the link between MS prognosis and social and territorial inequalities.

Exposure to sunlight is a known protective factor and is consistent with the north-east-south-west gradient observed in France. The choice of centers associated with the research, spread over the French territory, will make it possible to monitor and measure this effect in the prognosis of MS.

As the available treatments have evolved considerably over the last ten years, and in order to avoid a period effect, the patients recruited in the study will have to have a date of onset of the disease after 1 January 2009.

Primary objective Determining the relationship between socio-economic inequalities and the time to start disease-modifying therapy in MS Secondary objective

1. To determine the relationship between geographical inequalities and delay in starting disease-modifying therapy in MS
2. To determine the relationship between socio-economic inequalities and time to walking disability (EDSS 4)
3. To determine the relationship between geographical inequalities and time to walking disability (EDSS 4)
4. To measure the impact of disability on socioeconomic status in MS patients

ELIGIBILITY:
Inclusion criteria

* Be of legal age
* Have a confirmed MS according to the McDonald criteria 2017
* Have the date of onset of the disease recorded in EDMUS
* Have a disease onset date after 1 January 2009
* For patients receiving treatment for their MS*: have the date of first disease- modifying therapy entered in EDMUS

  * Patients not receiving treatment for their MS can be included if they meet the other criteria

Exclusion criteria

• Being deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population:
  Patients with a confirmed diagnosis of MS whose clinical data are present in the EDMUS database.
  Recruitment methods:
  Inclusion will be done during the usual consultations of the patients in their care centers, corresponding to one of the 4 investigating centers. The study will be offered to all patients who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-03-03 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The endpoint will be the time from disease onset to treatment, and the co-variates of the multivariate model will be all socio-demographic and clinical characteristics at disease onset. | The total time for a subject to participate is approximately 25 minutes, while reading the newsletter, asking questions if necessary and completing a questionnaire.
  The endpoint will be the time from disease onset to treatment, and the co-variates of the multivariate model will be all socio-demographic and clinical

SECONDARY OUTCOMES:
Delay before first treatment | The total time for a subject to participate is approximately 25 minutes, while reading the newsletter, asking questions if necessary and completing a questionnaire.
  Delay before first treatment
Time to reach an EDSS of more than 4 | The total time for a subject to participate is approximately 25 minutes, while reading the newsletter, asking questions if necessary and completing a questionnaire.
  Time to reach an EDSS of more than 4
Difference in disposable income between the start of the illness and the point date. | The total time for a subject to participate is approximately 25 minutes, while reading the newsletter, asking questions if necessary and completing a questionnaire.
  Difference in disposable income between the start of the illness and the point date.

CONTACTS AND LOCATIONS:
Overall Officials: Marc DEBOUVERIE, PU-PH, Principal Investigator — Service de Neurologie CHRU de Nancy; Aurélie RUET, PU-PH, Principal Investigator — Service de Neurologie et Maladies inflammatoires du systéme nerveux central; Gilles EDAN, PU-PH, Principal Investigator — PÔLE NEUROSCIENCES, CHU de Rennes; Pierre CLAVELOU, PU-PH, Principal Investigator — Service de Neurologie, CHU de Clermont-Ferrand
Locations (5):
- France (5):
  - Service de Neurologie et Maladies inflammatoires du Système nerveux central, Bordeaux
  - Service de Neurologie, Clermont-Ferrand
  - Service de Neurologie, Nancy
  - Pôle Neurosciences, Rennes
  - CIC 1433 Épidémiologie CliniqueInserm, CHRU, Université de Lorraine, Vandœuvre-lès-Nancy